CLINICAL TRIAL: NCT06064266
Title: Healthy Fat, Happy Microbiome (TAPIR), Proof-of-Concept Study
Acronym: TAPIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Mara van Trijp, PhD, Wageningen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL81345.081.23
Record Dates: First submitted 2023-09-12; First posted 2023-10-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Small Intestine
Keywords: Dietary fat; Microbial metabolites; Microbiota

STUDY DESIGN:
Intervention Model Description: 8-days preconditioning mild ketogenic controlled diet followed by a high fat shake challenge with a naso-intestinal catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8-days plant-based preconditioning mild ketogenic controlled diet followed by a high-fat shake. (Experimental)
  Interventions: Other: plant-based mild ketogenic controlled diet; Other: high-fat shake

INTERVENTIONS:
Other: plant-based mild ketogenic controlled diet — Plant-based mild ketogenic diet (10-20EN% carbohydrates, 10-20EN% protein, and 60-70EN% fat), consisting of a daily breakfast, lunch, dinner, and snacks.
Other: high-fat shake — The high-fat shake consists of unsweetened almond milk, sunflower oil, and plant sterols, resulting in a shake containing 885 kcal (1.5g protein, 97.3g fat, and 0.8g sugar).

SUMMARY:
Rationale: The role of dietary lipids in host-microbiome research has for a long time been overlooked; as high lipid intake has been recently indicated to have the most pronounced effect on the small intestinal microbiome, fecal-oriented studies might have missed their important, local effect. Indications for an interaction between dietary lipids and the small intestinal microbiome are mainly based on animal studies, but human data are largely missing. This study therefore aims at exploring this principal in vivo in healthy individuals.

Primary objective: To assess the effect of dietary lipids on the small intestinal microbiome in humans (proof-of-concept), the primary objective of our study is to measure production of microbiota-derived lipid metabolites in the human small intestine after consumption of a plant-based high-fat shake in healthy pre-conditioned subjects.

Secondary objectives: To explore future perspectives for dietary lipid - small intestinal microbiome interactive research, the secondary objectives of our study are

1. To compare the levels of microbiota-derived lipid metabolites in aspirate samples obtained through a naso-intestinal catheter (golden standard; invasive sampling method) and an aspiration capsule (less invasive, innovative sampling method), and in blood (local versus systemic effect) and feces (small intestinal versus fecal effect; less invasive sampling);
2. To investigate the acute effect of a high-fat shake on the composition and transcriptome activity of the small intestine microbiota in aspirate samples of healthy pre-conditioned subjects; 2a) To compare the acute effects on the small intestine microbiota composition in aspirate samples obtained through a naso-intestinal catheter versus those obtained via an aspiration capsule;
3. To study and compare the effect of a 8-day plant-based mild ketogenic preconditioning diet on the composition of the small intestine microbiota (aspiration capsule) and the fecal microbiota.

Study design: Proof-of-concept intervention study

Study population: 16 healthy adults, BMI between 18.5-30 kg/m2.

Intervention: 8-days preconditioning mild ketogenic controlled diet followed by a high fat shake challenge with a naso-intestinal catheter.

Main study parameters/endpoints: The primary study parameters are the microbial-derived metabolites from linoleic acid and plant sterols after consumption of the high fat shake.

Secondary study parameters include microbiota composition and transcriptome activity. Other parameters include inflammatory markers and ex-vivo analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* BMI 18.5-30 kg/m2
* Suitable veins for insertion of cannula

Exclusion Criteria:

* Having a history of medical or surgical events that may either put the subject at risk because of participation in the study, or influence the results of the study, including diabetes mellitus, dyslipidemia, a swallowing disorder, gastrointestinal or liver disease, irritable bowel syndrome, sleeping apnea, renal failure, cancer, nose/throat diseases, gastric bypass surgery, use of anticoagulants; as determined by the medical supervisor;
* Having a bleeding/coagulation disorder, including hemophilia, Von Willebrand disease, Bernard-Soulier, Glanzmann thrombasthenia or thrombocytopenia;
* Use of antibiotics within 3 months of starting the study or planned during the study;
* Use of any medications in the previous week that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, laxatives), or acidity (PPI, H2RA), as determined by medical supervisor;
* Use of pro- and prebiotic supplements within 4 weeks of starting the study;
* Planning or scheduled to undergo magnetic resonance imaging (MRI) at any time during the course of the study (the SIMBA Capsule is MR unsafe)
* Currently following a very low carbohydrate (ketogenic) diet;
* Having regularly less than 3 bowel movements per week (being constipated);
* Alcohol consumption >21 glasses a week (women) or >28 glasses a week (men);
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported);
* Not willing to give up blood donation during the study;
* Food allergies or intolerances for products that we use in the study;
* Current smokers;
* Current users of soft and/or hard drugs;
* Participation in another clinical trial at the same time;
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research or Human Nutrition and Health Department of Wageningen University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
lipid metabolites from linoleic acid and plant sterols in the small intestine aspirates | 0-6 hours
  Concentrations of microbiota-derived lipid metabolites in the small intestine aspirates, obtained by a naso-intestinal catheter, measured by lipidomics.

SECONDARY OUTCOMES:
lipid metabolites in small intestine aspirate samples obtained with an aspiration capsule. | 0-6 hours
  Concentrations of microbiota-derived lipid metabolites in the small intestine aspirates, obtained by an aspiration capsule, measured by lipidomics.
small intestine microbiota composition | 0-6 hours
  The relative composition (%) of the small intestine microbiota in aspirate samples obtained by an intestinal catheter.
small intestine microbiome capacity | 0-6 hours
  The functional capacity (transcriptomic activity) of the small intestine microbiota in aspirate samples obtained by an intestinal catheter.
Faecal microbiota | Baseline, after 8 days.
  The relative composition (%) of the faecal microbiota
Blood lipid metabolites | 0-6 hours
  Lipid metabolites (HYA, CLA, all untargeted lipid metabolites) will be measured in blood samples with lipidomics.
Blood triglycerides | 0-6 hours
  Concentrations of triglycerides
Blood free fatty acids | 0-6 hours
  Concentrations of free fatty acids
small intestine microbiota | Baseline, after 5 days.
  The relative composition (%) of the small intestine microbiota in aspirates obtained by an aspiration capsule.
small intestine microbiome | Baseline, after 5 days.
  The functional capacity (transcriptomic activity) of the small intestine microbiota in aspirates obtained by an aspiration capsule.

OTHER OUTCOMES:
Blood LPS | 0-6 hours
Blood ApoB48 | 0-6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] JanssenDuijghuijsen L, Fransen K, Deng R, Perenboom C, de Wit N, Hooiveld G, van Trijp M. How to Study the Effects of Dietary Lipids on the Small Intestinal Microbiome? Methodological Design and Evaluation of the Human HealThy fAt, haPpy mIcRobiome (TAPIR) Proof-of-Concept Study. Curr Dev Nutr. 2025 Feb 5;9(3):104564. doi: 10.1016/j.cdnut.2025.104564. eCollection 2025 Mar. PMID 40092654